CLINICAL TRIAL: NCT06436235
Title: Inflammation and Insulin Resistance in Kidney Stone Patients
Brief Title: Kidney Stone Inflammation
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB24-0024
Record Dates: First submitted 2024-05-03; First posted 2024-05-31 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Kidney Stone; Stone, Kidney
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Any urine or serum/plasma that is not utilized for the specified measurements in this study will be frozen at -80°C and retained as biospecimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kidney stone formers: The study team plans to enroll 20 non-diabetic participants with a history of at least one calcium-based kidney stone. Activities are the same for both cohorts, as follows:
  * Before clinic visit, participants will halt specific supplements and diuretics for a week.
  * At home, they complete a dietary questionnaire and collect 24-hour urine.
  * On the 7th day, they visit University of Chicago CRC. There, investigators will take measurements (height, weight) and DEXA scan, alongside kidney stone history review.
  * Throughout the day, participants provide urine and blood samples, undergo blood pressure checks, and fast until sample collection.
  * Samples undergo testing for kidney stone, inflammation, and diabetes risk factors and are stored for future research.
- Control cohort: The study team plans to enroll 20 healthy control participants with no history of kidney stones or family history of kidney stones. Activities are the same for both cohorts, as follows:
  * Before clinic visit, participants will halt specific supplements and diuretics for a week.
  * At home, they complete a dietary questionnaire and collect 24-hour urine.
  * On the 7th day, they visit University of Chicago CRC. There, investigators will take measurements (height, weight) and DEXA scan, alongside kidney stone history review.
  * Throughout the day, participants provide urine and blood samples, undergo blood pressure checks, and fast until sample collection.
  * Samples undergo testing for kidney stone, inflammation, and diabetes risk factors and are stored for future research.

SUMMARY:
This observational study aims to look at the connections between kidney stones, insulin resistance, and inflammation. The researchers hypothesize that people who form calcium kidney stones and have insulin resistance may have higher levels of inflammation because they have more visceral fat (fat around the abdominal organs).

The study will recruit 20 people who have had calcium kidney stones but don't have diabetes, and 20 healthy people who haven't had kidney stones. All the participants will come to the research center at the University of Chicago Medicine. Participants will have a dual-energy X-ray absorptiometry (DEXA) scan to measure their visceral fat, and give blood and urine samples. The blood will be tested for insulin resistance, inflammatory markers, and other metabolic factors. The urine will be analyzed for substances that increase kidney stone risk.

The main goal is to see if the kidney stone formers with insulin resistance have more visceral fat compared to those without insulin resistance and the healthy participants. The researchers will also compare inflammatory marker levels between groups, and look at how visceral fat, inflammatory markers, insulin resistance, and urine stone risk factors are related.

The findings may help explain how kidney stones are connected to metabolic conditions like diabetes and cardiovascular disease. Researchers hope this information will help identify stone formers at risk early and develop preventive treatments in the future.

DETAILED DESCRIPTION:
Participants will be recruited from the University of Chicago Medicine Kidney Stone Clinic (stone formers) and research participant registries (controls). After providing informed consent, participants will complete the following procedures:

Pre-Study:

1. One week prior, participants will discontinue vitamin C, multivitamins, calcium supplements, and diuretics.
2. One day prior, participants will complete a 24-hour urine collection and food frequency questionnaire at home.

Study Visit:

2. Participants will be admitted to the University of Chicago's Clinical Research Center (CRC) in a fasted state.

3. Three timed (45 minute) urine and blood specimen collections will occur.

4. Three seated blood pressure measurements will be taken.

5. Anthropometric measurements including height, weight, waist and neck circumference will be obtained.

6. A dual-energy X-ray absorptiometry (DEXA) scan will be performed to measure visceral fat content and bone density.

7. A brief clinical history will be obtained, including data on kidney stone episodes, procedures, and current stone burden.

8. Participants will remain fasted until all biological samples have been collected. Water intake will be allowed ad libitum.

Sample Analysis:

Urine:

1.24-hour and timed urine samples will be analyzed for kidney stone risk chemistries including volume, pH, solutes (calcium, oxalate, uric acid, citrate, etc).

2. Urine supersaturations for calcium oxalate, calcium phosphate, and uric acid will be calculated using EQUIL2 software.

3. Urine albumin and creatinine will be measured.

4. Remaining urine will be stored at -80°C for potential future assays.

Blood:

1. Serum glucose will be measured at the CRC laboratory.
2. Serum insulin, C-peptide, glucagon, GLP-1, and inflammatory markers (high-sensitivity CRP [C-reactive protein], IL-6, MMPs [matrix metalloproteinases], TNF-alpha, endotrophin) will be measured at the Diabetes Research and Training Center at the University of Chicago.
3. Other serum chemistries (electrolytes, calcium, creatinine, HbA1c, lipids) will be measured at the clinical laboratory.
4. Remaining serum will be stored at -80°C.

ELIGIBILITY:
Inclusion Criteria:

* Stone formers:
* Age 18-70
* History of at least one calcium-based kidney stone
* Healthy Controls:
* Age 18-70
* No history of kidney stone or family history of kidney stones

Exclusion Criteria (for both groups):

* History of primarily uric acid
* Cysteine, or struvite stones
* History of diabetes or impaired glucose tolerance
* Previous thiazide use
* Anyone on a medication that cannot be stopped that may affect urine composition
* Previous bariatric surgery or ileostomy
* Primary hyperparathyroidism and elevated serum calcium.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Kidney Stone Former Group:
  Age 18-70 years old History of at least one calcium-based kidney stone
  Control Group:
  Age 18-70 years old No personal history of kidney stones No family history of kidney stones
  Exclusion Criteria for Both Groups:
  History of primarily uric acid, cysteine, or struvite stones History of diabetes or impaired glucose tolerance Previous thiazide diuretic use Medications that cannot be stopped that may affect urine composition Previous bariatric surgery or ileostomy Primary hyperparathyroidism and elevated serum calcium
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Difference in visceral fat content in participants who form kidney stones with insulin resistance compared to participants who form kidney stones without insulin resistance and controls | 1 week total, one half day in the CRC
  Levels of visceral fat as measured by dual x-ray absorptiometry (DEXA).
Difference in inflammatory markers between participants who form kidney stones and controls | 1 week total, one half day in the CRC
  Markers of systemic inflammation, including high-sensitivity CRP, interleukin-6, MMP-7, MMP-9, TNF-alpha, and endotrophin.

SECONDARY OUTCOMES:
Correlation between visceral fat and inflammatory markers | 1 week total, one half day in the CRC
  Correlation between visceral fat levels (measured by dual x-ray absorptiometry [DEXA]) and the following markers of systemic inflammation:
  * High-sensitivity C-reactive protein (CRP)
  * Interleukin-6 (IL-6)
  * Matrix metalloproteinase-7 (MMP-7)
  * Matrix metalloproteinase-9 (MMP-9)
  * Tumor necrosis factor-alpha (TNF-alpha)
  * Endotrophin
Differences in urine composition | 1 week total, one half day in the CRC
  Differences in urine composition based on:
  * Levels of insulin resistance
  * Visceral fat content (measured by DEXA)
  * Levels of inflammatory markers (CRP, IL-6, MMP-7, MMP-9, TNF-alpha, endotrophin)
Differences in visceral fat levels | 1 week total, one half day in the CRC
  Differences in visceral fat levels (measured by DEXA) between kidney stone patients and controls
Differences in insulin resistance between kidney stone patients and controls | Time Frame: 1 week total, one half day in the CRC
  Differences in insulin resistance between kidney stone patients and controls, measured by:
  * Fasting blood glucose
  * Fasting insulin
  * Homeostatic model assessment of insulin resistance (HOMA-IR)
Differences in markers of systemic inflammation between kidney stone patients and controls | Time Frame: 1 week total, one half day in the CRC
  Differences in markers of systemic inflammation between kidney stone patients and controls, including:
  * High-sensitivity C-reactive protein (CRP)
  * Interleukin-6 (IL-6)
  * Matrix metalloproteinase-7 (MMP-7)
  * Matrix metalloproteinase-9 (MMP-9)
  * Tumor necrosis factor-alpha (TNF-alpha)
  * Endotrophin

CONTACTS AND LOCATIONS:
Overall Officials: Megan Prochaska, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States